CLINICAL TRIAL: NCT01080872
Title: Coronary Flow Reserve in Patients With Bio-active Stent or Everolimus-eluting Stent Implanted in Acute Coronary Syndrome
Acronym: BASE-CFR
Status: Completed | Type: Observational
Sponsor: The Hospital District of Satakunta (Other)
Responsible Party: Pasi Karjalainen, MD PhD, Satakunta Central Hospital
Other Study IDs: SA-005
Record Dates: First submitted 2010-03-03; First posted 2010-03-04 (Estimated); Last update posted 2011-05-05 (Estimated); Status verified 2011-05

CONDITIONS: Acute Coronary Syndrome
Keywords: acute coronary syndrome; coronary flow reserve; OCT; healing; drug eluting stent
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Titanium-NO coated stent: Patients receiving titanium-nitride-oxide coated stents during the intervention.
  Interventions: Device: CFR
- Everolimus eluting stent: Patients receiving everolimus eluting stents during the intervention.
  Interventions: Device: CFR

INTERVENTIONS:
Device: CFR — CFR will be assessed using transthoracic echocardiography with adenosine infusion.
  Other Names: Xience-V stent, Abbott vascular, USA

SUMMARY:
The aim of the trial is to assess coronary artery reactivity using adenosine-induced coronary flow reserve (CFR) by transthoracic echocardiography in patients with Bio-active stent (BAS) and Everolimus-eluting stent (EES) distal to the original culprit lesion at 6-8 months.

DETAILED DESCRIPTION:
Objective: The aim of the trial is to assess coronary artery reactivity using adenosine-induced coronary flow reserve (CFR) by transthoracic echocardiography in patients with Bio-active stent (BAS) and Everolimus-eluting stent (EES) distal to the original culprit lesion at 6-8 months.

Design: BASE-CFR is a substudy of the larger randomized multicenter BASE-ACS trial comparing bio-active Titan stent to everolimus-eluting stent in patients with acute coronary syndrome. CFR assessment will be performed at 6-8 months after stent implantation at the same time with OCT assessment. In-stent restenosis will be ruled out using OCT.

Primary endpoint: CFR at 6-8 months after stent implantation.

Secondary endpoint: Coronary flow velocity at baseline and during adenosine-induced hyperemia 6-8 months after stent implantation..

Association of CFR to unendotheliazed stent struts and stent malapposition.

Enrollment: 40 patients (20 receiving BAS and 20 receiving EES).

Clinical site: Satakunta Central Hospital, Finland Turku University Hospital, Finland

ELIGIBILITY:
Inclusion Criteria:

* The patient is enrolled to the BASE-ACS trial. Treated culprit lesion is in the proximal or middle LAD
* Patient or the patient's legal representative has been informed of the nature of the study and has provided written informed consent as approved by the Institutional Ethics Committee of the respective clinical site

Exclusion Criteria:

* Diabetes mellitus
* Treated stent position other than LAD proximal or middle.
* EF<30%
* Bifurcation lesions
* Renal impairment (creatinine >120 mmol/L)
* No suitable anatomy for OCT scan or CFR measurement

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute coronary syndrome who were treated with BAS or EES during index PCI.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Coronary flow reserve (CFR) | 6-8 months after stent implantation
  CFR at 6-8 months after stent implantation

SECONDARY OUTCOMES:
Coronary flow velocity | at baseline and during adenosine-induced hyperemia
Association of CFR to unendotheliazed stent struts and stent malapposition | 6-8 months

CONTACTS AND LOCATIONS:
Overall Officials: Tuomas O Kiviniemi, MD PhD, Study Chair — Satakunta Central Hospital; Antti Saraste, MD PhD, Study Chair — Turku University Hospital; Pasi P Karjalainen, MD PhD, Principal Investigator — Satakunta Central Hospital; Antti Ylitalo, MD PhD, Study Director — Satakunta Central Hospital; Jussi Mikkelsson, MD PhD, Study Chair — Satakunta Central Hospital
Locations (2):
- Finland (2):
  - Satakunta Central Hospital, Pori
  - Turku University Hospital, Turku

REFERENCES:
- [Background] Kiviniemi T. Assessment of coronary blood flow and the reactivity of the microcirculation non-invasively with transthoracic echocardiography. Clin Physiol Funct Imaging. 2008 May;28(3):145-55. doi: 10.1111/j.1475-097X.2008.00794.x. Epub 2008 Feb 26. PMID 18312446
- [Derived] Karjalainen P, Kiviniemi TO, Lehtinen T, Nammas W, Ylitalo A, Saraste A, Mikkelsson J, Pietila M, Biancari F, Airaksinen JK. Neointimal coverage and vasodilator response to titanium-nitride-oxide-coated bioactive stents and everolimus-eluting stents in patients with acute coronary syndrome: insights from the BASE-ACS trial. Int J Cardiovasc Imaging. 2013 Dec;29(8):1693-703. doi: 10.1007/s10554-013-0285-8. Epub 2013 Aug 31. PMID 23996244